CLINICAL TRIAL: NCT01360437
Title: Ticagrelor in Comparison to Prasugrel for Inhibition of Platelet Reactivity, in Patients With Acute Coronary Syndrome (ACS) Presenting Resistance to the Usual Clopidogrel Dose After PCI
Brief Title: Ticagrelor Versus Prasugrel in Acute Coronary Syndromes After Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-6
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: coronary angioplasty; clopidogrel hyporesponsiveness; prasugrel; ticagrelor; CAD; ACS
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator)
  Interventions: Drug: Prasugrel
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10mg/day
  Arms: Prasugrel
Drug: Ticagrelor — Ticagrelor 90mg twice a day
  Arms: Ticagrelor

SUMMARY:
This is a single-center, randomized, single-blind, investigator-initiated pharmacological study with a crossover design. Patients with acute coronary syndrome (ST-elevation myocardial infarction, non-ST elevation myocardial infarction, unstable angina) and presenting high on-clopidogrel platelet reactivity as assessed with the VerifyNow assay (platelet reactivity units PRU≥235) 24 hours post percutaneous coronary intervention (PCI), will be randomized after informed consent in a 1:1 ratio to either prasugrel 10mg/d or ticagrelor 90mg twice a day for 15 days. Platelet reactivity assessment will be performed at Day 15±2 days and then a crossover directly to the alternate treatment group for an additional 15 days period, without an intervening washout period will be carried out. Patients will return at Day 30±2 days for platelet reactivity assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients having PCI with stenting 24 hours prior randomization, meeting one of the following criteria :

   * Acute coronary syndrome (unstable angina or myocardial infarction)
   * TIMI risk score>2
3. Platelet reactivity in PRU ≥235 24 hours post-PCI
4. Informed consent obtained in writing

Exclusion Criteria:

* Treatment with other investigational agents (including placebo) or devices within 30 days prior to randomization or planned use of investigational agents or devices prior to the Day 30 visit.
* Pregnancy
* Breastfeeding
* Inability to give informed consent or high likelihood of being unavailable for the Day 30 follow up.
* Prior PCI performed within 30 days prior to randomization
* Cardiogenic shock
* Major periprocedural complications (death, stent thrombosis, vessel perforation, arrhythmias requiring cardioversion, temporary pacemaker insertion or intravenous antiarrhythmic agents, respiratory failure requiring intubation, vascular injury (pseudoaneurysm, arteriovenous shunt, retroperitoneal bleeding or hematoma >5 cm at the arterial catheter insertion site), major bleeding (need for bood transfusion or drop in haemoglobin post-PCI by ≥ 5 gr/ dl or intracranial bleeding).
* Unsuccessful PCI (residual stenosis > 30% or flow < ΤΙΜΙ 3) or planned staged PCI in the next 30 days after randomization
* Requirement for oral anticoagulant prior to the Day 30 visit
* Current or planned therapy with other thienopyridine class of ADP receptor inhibitors.
* Known hypersensitivity to prasugrel or ticagrelor
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding on longterm thienopyridine therapy.
* Any previous history of ischemic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
* Thombocytopenia (<100.000 / μL) at randomization
* Anaemia (Hct <30%) at randomization
* Polycytaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitors administration
* Severe allergy to contrast agent, unfractionated heparin, enoxaparin or bivalirudin that cannot be adequately premedicated.
* Recent (< 6 weeks) major surgery or trauma, including GABG.
* Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardiac events.
* Dialysis required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity Units (PRU) assessed by VerifyNow (Accumetrics) | Day 15
  The primary outcome will be assessed 15 days after the onset of each study drug

SECONDARY OUTCOMES:
Hyporesponsiveness rate (PRU≥235) at the end of the 2 treatment periods | Day 15
  Hyporesponsiveness rate will be assessed 15 days after the onset of each study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Patras University Hospital, Rio, Patras, Greece

REFERENCES:
- [Derived] Alexopoulos D, Galati A, Xanthopoulou I, Mavronasiou E, Kassimis G, Theodoropoulos KC, Makris G, Damelou A, Tsigkas G, Hahalis G, Davlouros P. Ticagrelor versus prasugrel in acute coronary syndrome patients with high on-clopidogrel platelet reactivity following percutaneous coronary intervention: a pharmacodynamic study. J Am Coll Cardiol. 2012 Jul 17;60(3):193-9. doi: 10.1016/j.jacc.2012.03.050. PMID 22789884